CLINICAL TRIAL: NCT04232176
Title: Precision of Optical Diagnosis in Polyps Between 5-15 mm and Its Implications on Surveillance. A Prospective, Multicenter Study.
Acronym: POPS
Status: Completed | Type: Observational
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, EDUARDO REDONDO CEREZO, MD, PhD, Head of Gastroenterology, University Hospital Virgen de las Nieves
Other Study IDs: POPS.HUVN.19
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Colonic Polyps; Colon Neoplasms; Colon Cancer; Serrated Adenoma
Keywords: Endoscopic optical diagnosis
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the ability of endoscopists to perform a complete optical diagnosis of colorectal polyps between 5 and 15 mm, and the impact of the only endoscopic diagnosis on the follow-up program for those patients. This is a prospective study in which we compare the diagnosis regarding size and histology made by the endoscopist versus de pathologic diagnosis.

DETAILED DESCRIPTION:
Background: Optical diagnosis of colonic polyps is an attractive possibility and a common practice. However, recommendations and the main decision concerning patients' management still rely on histological diagnosis, with controversial results in previous studies, usually designed to analyze the accuracy of this diagnosis in the setting of a 'resect and discard' or 'diagnose and leave' strategy. However, little has been studied on this diagnosis on polyps of about 10 mm, the threshold for the consideration as a high risk adenoma, that need a 3 year colonoscopy, or, in case of a smaller adenoma, with a recommended revision in 5 years. Some studies have addressed the accuracy when estimating the polyp size, and others the histology by means of virtual or optical chromoendoscopy, but no one has studied both parameters, that are the two pillars in which a revision program for the patient is decided.

Hypothesis: Our main purpose is to determine the accuracy of the complete optical diagnosis as made by the endoscopist in the endoscopy room, in order to give recommendations immediately after the colonoscopy, with no need of further histological analyses.

Aims:

* To establish endoscopist accuracy, in different hospital settings, to predict size and histology of polyps between 5 and 15 mm and whether follow-up recommedations based on this diagnosis are accurate enough, when compared to the pathologic diagnosis.
* To evaluate accuracy of the optical size estimation by the endoscopist, with respect to the measurement after resection and by the pathologist (after formaline fixation).
* To analyze the rate of sessile serrated adenoma not diagnosed by the endoscopista on site.
* To determine the proportion of incomplete resection and complications with different resection techniques.
* To follow-up patients with high risk adenoma with the aim to establish the best follow-up schedule for those patients, and clarify this topic, still subjected to uncertainty.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years
* Colorectal polyps with an estimated size (endoscopist estimation) between 5 and 15 mm.
* Consent to be included in the protocol.

Exclusion Criteria:

* Polyps sized <5 mm or >15 mm
* Polyps that cannot be resected.
* Polys that cannot be sent for pathologic study.
* Peacemeal resection.
* Polyposis syndromes with a previous histologic diagnosis.
* Patients do not consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that come to the endoscopy unit for colorectal cancer screening or with a specific clinical indication during the study period, in any of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Concordance of optical diagnosis with pathologic diagnosis | Immediate after the polyps detection
  Optical diagnosis accuracy (endoscopist) when compared to the Pathologic report
Precision in polyps sizing the pathologist | Immediate after resection and within 10 days after polyp resection to allow pathologic diagnosis
  Comparison of sizes after resection and after formaline and pathologic diagnosis

SECONDARY OUTCOMES:
Rate of polyps' recurrence at the end of the follow-up. | 5 years after the index resection
  Polyps recurrence after long-term follow up for advanced adenoma (Rate)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Heredia-Carrasco, MD, Principal Investigator — 'Virgen de las Nieves' University Hospital. Granada
Locations (1):
- "Virgen de las Nieves" University Hospital, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heitman SJ, Ronksley PE, Hilsden RJ, Manns BJ, Rostom A, Hemmelgarn BR. Prevalence of adenomas and colorectal cancer in average risk individuals: a systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1272-8. doi: 10.1016/j.cgh.2009.05.032. Epub 2009 Jun 10. PMID 19523536
- [Background] Butterly LF, Chase MP, Pohl H, Fiarman GS. Prevalence of clinically important histology in small adenomas. Clin Gastroenterol Hepatol. 2006 Mar;4(3):343-8. doi: 10.1016/j.cgh.2005.12.021. PMID 16527698
- [Background] Mason SE, Poynter L, Takats Z, Darzi A, Kinross JM. Optical Technologies for Endoscopic Real-Time Histologic Assessment of Colorectal Polyps: A Meta-Analysis. Am J Gastroenterol. 2019 Aug;114(8):1219-1230. doi: 10.14309/ajg.0000000000000156. PMID 30848728
- [Background] Rex DK, Kahi C, O'Brien M, Levin TR, Pohl H, Rastogi A, Burgart L, Imperiale T, Ladabaum U, Cohen J, Lieberman DA. The American Society for Gastrointestinal Endoscopy PIVI (Preservation and Incorporation of Valuable Endoscopic Innovations) on real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2011 Mar;73(3):419-22. doi: 10.1016/j.gie.2011.01.023. PMID 21353837
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] McGill SK, Evangelou E, Ioannidis JP, Soetikno RM, Kaltenbach T. Narrow band imaging to differentiate neoplastic and non-neoplastic colorectal polyps in real time: a meta-analysis of diagnostic operating characteristics. Gut. 2013 Dec;62(12):1704-13. doi: 10.1136/gutjnl-2012-303965. Epub 2013 Jan 7. PMID 23300139
- [Background] IJspeert JE, Bastiaansen BA, van Leerdam ME, Meijer GA, van Eeden S, Sanduleanu S, Schoon EJ, Bisseling TM, Spaander MC, van Lelyveld N, Bargeman M, Wang J, Dekker E; Dutch Workgroup serrAted polypS & Polyposis (WASP). Development and validation of the WASP classification system for optical diagnosis of adenomas, hyperplastic polyps and sessile serrated adenomas/polyps. Gut. 2016 Jun;65(6):963-70. doi: 10.1136/gutjnl-2014-308411. Epub 2015 Mar 9. PMID 25753029
- [Background] Iacucci M, Trovato C, Daperno M, Akinola O, Greenwald D, Gross SA, Hoffman A, Lee J, Lethebe BC, Lowerison M, Nayor J, Neumann H, Rath T, Sanduleanu S, Sharma P, Kiesslich R, Ghosh S, Saltzman JR; SIMPLE classification investigator team. Development and validation of the SIMPLE endoscopic classification of diminutive and small colorectal polyps. Endoscopy. 2018 Aug;50(8):779-789. doi: 10.1055/s-0044-100791. Epub 2018 Mar 23. PMID 29571175
- [Background] Izzy M, Virk MA, Saund A, Tejada J, Kargoli F, Anand S. Accuracy of endoscopists' estimate of polyp size: A continuous dilemma. World J Gastrointest Endosc. 2015 Jul 10;7(8):824-9. doi: 10.4253/wjge.v7.i8.824. PMID 26191348
- [Background] Rees CJ, Rajasekhar PT, Wilson A, Close H, Rutter MD, Saunders BP, East JE, Maier R, Moorghen M, Muhammad U, Hancock H, Jayaprakash A, MacDonald C, Ramadas A, Dhar A, Mason JM. Narrow band imaging optical diagnosis of small colorectal polyps in routine clinical practice: the Detect Inspect Characterise Resect and Discard 2 (DISCARD 2) study. Gut. 2017 May;66(5):887-895. doi: 10.1136/gutjnl-2015-310584. Epub 2016 Apr 19. PMID 27196576
- [Derived] Redondo-Cerezo E, Heredia-Carrasco C, Alegria-Motte C, Caballero-Mateos A, Vadillo-Calles F, Ortega-Suazo EJ, Martos-Ruiz V, Ariza-Fernandez JL, Lopez-Gonzalez E, Martinez-Cara JG, Valverde-Lopez F, de Hierro ML, Sanchez-Capilla D, Lopez-Hidalgo JL, Jimenez-Rosales R. Accuracy in optical diagnosis for polyps between 5 and 15 mm and its implications on surveillance. A prospective, multicenter study. (POPS study). Surg Endosc. 2022 Jul;36(7):5356-5365. doi: 10.1007/s00464-021-08917-w. Epub 2022 Jan 6. PMID 34988735